CLINICAL TRIAL: NCT05020236
Title: AN OPEN-LABEL, 3-ARM, MULTICENTER, RANDOMIZED PHASE 3 STUDY TO EVALUATE THE EFFICACY AND SAFETY OF ELRANATAMAB (PF-06863135) MONOTHERAPY AND ELRANATAMAB + DARATUMUMAB VERSUS DARATUMUMAB + POMALIDOMIDE + DEXAMETHASONE IN PARTICIPANTS WITH RELAPSED/REFRACTORY MULTIPLE MYELOMA WHO HAVE RECEIVED AT LEAST 1 PRIOR LINE OF THERAPY INCLUDING LENALIDOMIDE AND A PROTEASOME INHIBITOR
Brief Title: A Study to Learn About the Study Medicine Elranatamab Alone and With Daratumumab in People With Multiple Myeloma Who Have Received Other Treatments
Acronym: MAGNETISMM-5
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: C1071005; MAGNETISMM-5 (Other: Alias Study Number); 2023-509208-14-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2021-08-11; First posted 2021-08-25 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Elranatamab; PF-06863135; B-Cell Maturation Antigen; BCMA; Bispecific antibody; BCMA-CD3 bispecific antibody; Daratumumab; Pomalidomide; Multiple myeloma; Relapsed multiple myeloma; Refractory multiple myeloma; MagnetisMM-5
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Injections; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1 Safety Lead-In Dose Escalation: Elranatamab + Daratumumab (Experimental)
  Interventions: Drug: Elranatamab; Drug: Daratumumab
- Part 2 Randomized Arm A: Elranatamab (Experimental)
  Interventions: Drug: Elranatamab
- Part 2 Randomized Arm B: Elranatamab + Daratumumab (Experimental)
  Interventions: Drug: Elranatamab; Drug: Daratumumab
- Part 2 Randomized Arm C: Daratumumab + Pomalidomide + Dexamethasone (Active Comparator)
  Interventions: Drug: Daratumumab; Drug: Pomalidomide; Drug: Dexamethasone
- Part 3 Arm D: Elranatamab (Experimental)
  Interventions: Drug: Elranatamab
- Part 3 Arm E: Elranatamab + Daratumumab (Experimental)
  Interventions: Drug: Elranatamab; Drug: Daratumumab

INTERVENTIONS:
Drug: Elranatamab — subcutaneous
  Other Names: PF-06863135
  Arms: Part 1 Safety Lead-In Dose Escalation: Elranatamab + Daratumumab; Part 2 Randomized Arm A: Elranatamab; Part 2 Randomized Arm B: Elranatamab + Daratumumab; Part 3 Arm D: Elranatamab; Part 3 Arm E: Elranatamab + Daratumumab
Drug: Daratumumab — Daratumumab / hyaluronidase, subcutaneous
  Other Names: Darzalex Faspro; Darzalex solution for injection
  Arms: Part 1 Safety Lead-In Dose Escalation: Elranatamab + Daratumumab; Part 2 Randomized Arm B: Elranatamab + Daratumumab; Part 2 Randomized Arm C: Daratumumab + Pomalidomide + Dexamethasone; Part 3 Arm E: Elranatamab + Daratumumab
Drug: Pomalidomide — oral
  Other Names: Pomalyst, Imnovid
  Arms: Part 2 Randomized Arm C: Daratumumab + Pomalidomide + Dexamethasone
Drug: Dexamethasone — oral
  Arms: Part 2 Randomized Arm C: Daratumumab + Pomalidomide + Dexamethasone

SUMMARY:
The purpose of this clinical trial is to (1) learn whether the BCMA-CD3 bispecific antibody elranatamab can provide more benefit to people with multiple myeloma compared to a combination therapy including daratumumab, pomalidomide, and dexamethasone, and (2) learn about the safety and activity of elranatamab in combination with the anti-CD38 monoclonal antibody daratumumab. People with multiple myeloma who have received previous treatment including lenalidomide will be enrolled in the study.

Part 1 of the study will assess the safety and activity of different doses of elranatamab in combination with daratumumab.

People participating in Part 2 of the study will be randomly assigned to receive either elranatamab alone, elranatamab plus daratumumab, or daratumumab, pomalidomide, and dexamethasone. Part 2 will evaluate the safety and activity of (1) elranatamab alone compared to daratumumab, pomalidomide, and dexamethasone, and (2) elranatamab plus daratumumab.

Part 3 will assess the effect of increased measures to protect against infection in people treated with either elranatamab alone or together with daratumumab.

All people participating in the study will receive study treatment until their disease progresses, they experience unacceptable side effects, or they choose to no longer participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of multiple myeloma as defined by IMWG criteria (Rajkumar et al, 2014).
* Measurable disease based on IMWG criteria as defined by at least 1 of the following:

  * Serum M-protein ≥0.5 g/dL.
  * Urinary M-protein excretion ≥200 mg/24 hours.
  * Serum immunoglobulin FLC ≥10 mg/dL (≥100 mg/L) AND abnormal serum immunoglobulin kappa to lambda FLC ratio (<0.26 or >1.65).
* Prior anti-multiple myeloma therapy including treatment with lenalidomide.
* ECOG performance status ≤2.
* Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade ≤1.
* Not pregnant and willing to use contraception.

Exclusion Criteria:

* Smoldering multiple myeloma.
* Plasma cell leukemia.
* Amyloidosis.
* POEMS Syndrome.
* Stem cell transplant within 12 weeks prior to enrolment, or active graft versus host disease.
* Active HBV, HCV, SARS-CoV2, HIV, or any active, uncontrolled bacterial, fungal, or viral infection.
* Any other active malignancy within 3 years prior to enrolment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ.
* Previous treatment with a BCMA-directed therapy.
* Live attenuated vaccine within 4 weeks of the first dose of study intervention.
* Administration with an investigational product (e.g. drug or vaccine) concurrent with study intervention or within 30 days preceding the first dose of study intervention used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 944 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2026-04-27 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Part 1 Safety Lead-In: Incidence of dose limiting toxicities | First 42 days after first elranatamab dose
Part 2 Randomized: Progression free survival per International Myeloma Working Group criteria | From date of randomization to date of progressive disease, discontinuation from the study, death, or censoring, whichever occurs first, assessed up to 51 months
Part 3: Frequency of treatment-emergent adverse events | First 84 days after first elranatamab dose

SECONDARY OUTCOMES:
Part 1 Safety Lead-In: Progression free survival per International Myeloma Working Group criteria | From date of randomization to date of progressive disease, discontinuation from study, death, or censoring, whichever occurs first, assessed up to 51 months
Overall survival | From date of randomization to date of discontinuation from study, death, or censoring, whichever occurs first, assessed up to 51 months
Objective response rate per International Myeloma Working Group criteria | From date of randomization to date of progressive disease, discontinuation from study, death, or start of new anticancer therapy, whichever occurs first, assessed up to 51 months
Duration of response per International Myeloma Working Group criteria | From date of confirmed objective response to date of progressive disease, discontinuation from study, death, or censoring, whichever occurs first, assessed up to 51 months
Time to response per International Myeloma Working Group criteria | From date of randomization to date of confirmed objective response, assessed up to 51 months
Complete response rate per International Myeloma Working Group criteria | From date of randomization to date of progressive disease, discontinuation from study, death, or start of new anticancer therapy, whichever occurs first, assessed up to 51 months
Duration of complete response per International Myeloma Working Group criteria | From date of confirmed complete response to date of progressive disease, discontinuation from study, death, or censoring, whichever occurs first, assessed up to 51 months
Minimal residual disease negativity rate per International Myeloma Working Group criteria | From date of randomization to date of progressive disease, discontinuation from study, death, or start of new anticancer therapy, whichever occurs first, assessed up to 51 months
Sustained minimal residual disease negativity rate per International Myeloma Working Group criteria | From date of randomization to date of progressive disease, discontinuation from study, death, or start of new anticancer therapy, whichever occurs first, assessed up to 51 months
Progression free survival on next-line treatment per International Myeloma Working Group criteria | From date of randomization to date of second objective disease progression, discontinuation from the study, death, or censoring, whichever occurs first, assessed up to 51 months
Frequency of treatment-emergent adverse events | From date of first dose of study intervention through minimum of 90 days after last study intervention administration. Reporting of non-serious AEs ends at start of new anti-cancer therapy.
Frequency of abnormal laboratory results | From date of first dose of study intervention through minimum of 90 days after last study intervention administration. Reporting of non-serious AEs ends at start of new anti-cancer therapy.
Rate of Grade ≥2 cytokine release syndrome | First 28 days after first elranatamab dose
Elranatamab pharmacokinetics by pre- and post-dose concentrations | From date of first dose through up to 14 days after date of last dose of elranatamab
Elranatamab immunogenicity by anti-drug antibodies against elranatamab | From date of first dose through up to 14 days after date of last dose of elranatamab
Daratumumab pharmacokinetics by pre-dose concentrations | From date of first dose through up to 14 days after date of last dose of daratumumab
Health-related quality of life by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 | From date of informed consent through up to 35 days after date of last dose of study intervention
Health-related quality of life by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Myeloma 20 | From date of informed consent through up to 35 days after date of last dose of study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (238):
- United States (27):
  - Clovis Community Medical Center, Clovis, California
  - Community Cancer Institute, Clovis, California
  - University of California San Francisco, Fresno, California
  - Community Regional Medical Center, Fresno, California
  - UCHealth Poudre Valley Hospital, Fort Collins, Colorado
  - UCHealth Harmony, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth - Medical Center of the Rockies, Loveland, Colorado
  - Sylvester Comprehensive Cancer Center - Aventura, Aventura, Florida
  - Sylvester Comprehensive Cancer Center- The Lennar Foundation Medical Center, Coral Gables, Florida
  - Sylvester Comprehensive Cancer Center - Coral Springs, Coral Springs, Florida
  - University of Miami Hospital and Clinics - Deerfield Beach, Deerfield Beach, Florida
  - Sylvester Comprehensive Cancer Center - Hollywood, Hollywood, Florida
  - Griffin Cancer Research Building (GCRB), Miami, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Miami Hospital and Clinics, Miami, Florida
  - Sylvester Comprehensive Cancer Center - Kendall, Miami, Florida
  - Sylvester Comprehensive Cancer Center - Plantation, Plantation, Florida
  - East Jefferson General Hospital, Metairie, Louisiana
  - MSK Basking Ridge, Basking Ridge, New Jersey
  - MSK Monmouth, Middletown, New Jersey
  - MSK Bergen, Montvale, New Jersey
  - MSK Commack, Commack, New York
  - MSK Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center - David H. Koch Center for Cancer Care (74th Street)., New York, New York
  - Memorial Sloan Kettering Cancer Center - Main Campus, New York, New York
  - MSK Nassau, Uniondale, New York
- Argentina (7):
  - Alexander Fleming S.A (Instituto Medico Especializado Alexander Fleming), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - FUNDALEU - Fundacion para combatir la Leucemia, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - FUNDALEU -Fundación para combatir la leucemia, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - FUNDALEU, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - Hospital Universitario Austral, Presidente Derqui, Buenos Aires
  - Sanatorio de La Mujer, Rosario, Santa Fe Province
- Australia (12):
  - Pindara Private Hospital, Benowa, Queensland
  - QScan Radiology Clinics, Clayfield, Queensland
  - Gallipoli Medical Research Foundation, Greenslopes, Queensland
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Epworth Freemasons, East Melbourne, Victoria
  - St Vincent's Hospital (Melbourne), Fitzroy, Victoria
  - Barwon Health, Geelong, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Epworth Healthcare, Richmond, Victoria
  - Slade Pharmacy, Richmond, Victoria
  - Linear Clinical Research, Perth, Western Australia
- Austria (5):
  - Universitätsklinikum Krems, Krems, Lower Austria
  - Klinik Ottakring, Vienna, Vienna
  - Universitätsklinik für Innere Medizin V Innsbruck, Innsbruck
  - Uniklinikum Salzburg, Salzburg
  - Medizinische Universität Wien, Vienna
- Belgium (2):
  - Grand Hôpital de Charleroi, Gilly, Hainaut
  - CHU UCL Namur (site Godinne), Yvoir, Namur
- Brazil (14):
  - Instituto D'Or de Pesquisa e Ensino (IDOR) - Filial Salvador, Salvador, Estado de Bahia
  - Centro Gaucho Integrado De Oncologia, Hematologia, Ensino E Pesquisa, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Clínica - Área Administrativa, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - BP - A Beneficencia Portuguesa de São Paulo, São Paulo, São Paulo
  - Clínica Médica São Germano LTDA, SP, São Paulo
  - Hospital Américas Medical City, Rio de Janeiro
  - Instituto de Educação, Pesquisa e Gestão em Saúde, Rio de Janeiro
  - ESHO Empresa de Serviços Hospitalares S.A/ Hospital Samaritano de Higienópolis, São Paulo
  - IDOR Ensino e Pesquisa, São Paulo
  - HU UNIFESP / SPDM - Hospital São Paulo, São Paulo
  - Universidade Federal de Sao Paulo, São Paulo
  - Clínica Médica São Germano S/S Ltda, São Paulo
  - Instituto D'Or de Pesquisa e Ensino (IDOR), São Paulo
- Canada (9):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - QEII Health Sciences Centre - Victoria General Site, Halifax, Nova Scotia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Hamilton Health Sciences-Juravinski Cancer Centre, Hamilton, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CIUSSS de l'Est-de-l'Île-de-Montréal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Saskatoon Cancer Center, Saskatoon, Saskatchewan
- China (22):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Nanjing Drum Tower Hospital ， The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Province Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shandong Provincial Hospital, Jinan, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Institute of hematology&blood disease hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Beijing Boren Hospital, Beijing
  - Chongqing University Cancer Hospital, Chongqing
- Czechia (7):
  - Fakultní nemocnice Brno Bohunice, Brno, Brno-m?sto
  - Fakultni Nemocnice Plzen, Plzen - Lochotin, Plzeň Region
  - Fakultni poliklinika, Prague, Praha 2
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Ostrava, Ostrava-Poruba
  - Vseobecna fakultni nemocnice v Praze, Prague
- Finland (6):
  - Kuopion Yliopistollinen Sairaala, Kuopio, Northern Savonia
  - Tampereen yliopistollinen sairaala, Tampere, Pirkanmaa
  - Turku University Hospital, Turku, Southwest Finland
  - Helsinki University Hospital - Comprehensive Cancer Center (HYKS - Syöpäkeskus), Helsinki
  - Oulun yliopistollinen sairaala, Oulu
  - Tampereen yliopistollinen sairaala, Tampere
- France (8):
  - Centre Hospitalier Universitaire de Limoges - Hôpital Dupuytren, Limoges, Limousin
  - Hopital Claude Huriez - CHU de Lille, Lille, NORD
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu, Nantes
  - Hopital Necker, Paris
  - Hôpital Saint Antoine, Paris
  - Centre Hospitalier Lyon Sud - Service d'Hematologie Clinique, Pierre-Bénite
  - CHU de Poitiers, Hôpital de la Milétrie, Pôle Régional de Cancérologie, Poitiers
  - Institut Universitaire du Cancer Toulouse - Oncopole - CHU de TOULOUSE, Toulouse
- Germany (6):
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Charité Universitätsmedizin Berlin, Berlin
  - Staedtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Klinikum Chemnitz gGMbH, Chemnitz
  - Universitätsklinikum rechts der Isar, Technische Universität München (TUM), München
- Greece (5):
  - Evangelismos General Hospital of Athens, Athens, Attikí
  - Radiology vendor, Athens, Attikí
  - Alexandra General Hospital of Athens, Athens, Attikí
  - Theageneio Cancer Hospital of Thessaloniki, Thessaloniki, Kentrikí Makedonía
  - University General Hospital of Ioannina, Ioannina
- Italy (9):
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori", Meldola, Emilia-Romagna
  - Ospedale San Martino, Genoa, Liguria
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Lombardy
  - ASST Santi Paolo e Carlo Ospedale San Carlo Borromeo SSD di Onco-Ematologia (Edificio C-piano terra), Milan, Milan
  - Policlinico "G. Rodolico", Catania, Sicily
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna
  - AOU Policlinico Umberto I, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
- Japan (16):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - University of Fukui Hospital, Yoshida-gun, Fukui
  - National Hospital Organization Shibukawa Medical Center, Shibukawa, Gunma
  - Iwate Medical University Hospital, Yahaba-cho, Iwate
  - Tohoku University Hospital, Sendai, Miyagi
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Japanese Red Cross Medical Center, Shibuya-ku, Tokyo
  - Akita University Hospital, Akita
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kagoshima University Hospital, Kagoshima
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Nagasaki University Hospital, Nagasaki
  - National Hospital Organization Okayama Medical Center, Okayama
  - Osaka Metropolitan University Hospital, Osaka
  - Tokushima University Hospital, Tokushima
  - Yamagata University Hospital, Yamagata
- Mexico (4):
  - Hematológica Alta Especialidad SC, consultorio 830, Colonia Valle de Las Palmas, México
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City
  - Instituto Veracruzano en Investigación Clínica S.C., Veracruz
- Netherlands (2):
  - Erasmus Universitair Medisch Centrum, Rotterdam, South Holland
  - Maastricht University Medical Center, Maastricht
- New Zealand (10):
  - North Shore Hospital, Auckland
  - Labtests Auckland Ltd., Auckland
  - Aotearoa Clinical Trials, Auckland
  - Waikato District Health Board, Waikato Hospital, Hamilton
  - TRG Imaging, Milford
  - Pacific Radiology, Newtown
  - Broadway Radiology, Palmerston North
  - Palmerston North Hospital, Roslyn
  - Pharmacy on Shakespeare, Takapuna
  - Capital, Coast and Hutt Valley District - Wellington Regional Hospital, Wellington
- Norway (4):
  - Haukeland Universitetssjukehus, Bergen, Hordaland
  - Stavanger Universitetssykehus, Stavanger, Rogaland
  - Oslo Universitetssykehus Ullevål, Oslo
  - St Olavs Hospital, Trondheim
- Poland (7):
  - Szpital Uniwersytecki nr 2 im. dr Jana Biziela w Bydgoszczy Klinika Hematologii, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Pratia Onkologia Katowice, Katowice
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Centrum Medyczne Pratia Poznan, Skorzewo
  - Uniwersyteckie Centrum Kliniczne WUM Centralny Szpital Kliniczny, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw
- South Korea (9):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeonranamdo
  - Pusan National University Hospital, Busan, Pusan-kwangyǒkshi
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Kyungpook National University Hospital, Daegu, Taegu-kwangyǒkshi
  - Gachon University Gil Medical Center, Incheon
  - Asan Medical Center, Seoul
- Spain (14):
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruna
  - Institut Català d'Oncologia - L'Hospitalet, L'Hospitalet Del Llobregat, Barcelona [barcelona]
  - Hospital Universitari Mutua Terrassa, Terrassa, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario de Toledo, Toledo, Other
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitari De Girona Doctor Josep Trueta, Girona
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitario y Politecnico La Fe, Valencia
- Sweden (8):
  - Skånes Universitetssjukhus Lund, Lund, Skåne LÄN [se-12]
  - Södra Älvsborg Sjukhus, Borås
  - Falu Lasarett, Falun
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Sunderby Sjukhus, Luleå
  - Universitetssjukhuset Örebro, Örebro, Örebro LÄN [se-18]
  - Läkemedelsberedningen, Linköping, Östergötlands LÄN [se-05]
  - Universitetssjukhuset i Linköping, Linköping, Östergötlands LÄN [se-05]
- Taiwan (5):
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (14):
  - Istanbul Universitesi Istanbul Tıp Fakultesi Hastanesi, Istanbul, İ̇stanbul
  - Medipol Mega Universite Hastanesi, Istanbul, İ̇stanbul
  - Acibadem Universitesi Atakent Hastanesi, Istanbul, İ̇stanbul
  - Sisli Florence Nightingale Hastanesi, Istanbul, İ̇stanbul
  - Ege Universitesi Hastanesi, Izmir, İ̇zmir
  - Dokuz Eylul Universitesi Hastanesi, Izmir, İ̇zmir
  - Baskent Universitesi Adana Dr. Turgut Noyan Uygulama ve Arastirma Merkezi, Adana
  - Ankara University Health Practice and Research Hospitals, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastırma Hastanesi, Ankara
  - Akdeniz Universitesi Hastanesi, Antalya
  - Gaziantep Universitesi Sahinbey Arastirma ve Uygulama Hastanesi, Gaziantep
  - Erciyes Universitesi Tıp Fakultesi Hastaneleri, Kayseri
  - Özel Anadolu Sağlık Merkezi, Kocaeli
  - Inonu Universitesi Turgut Ozal Tıp Merkezi, Malatya
- United Kingdom (6):
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - Churchill Hospital, Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire
  - University Hospital of Wales, Cardiff, South Glamorgan
  - Bristol Haematology and Oncology Centre, Bristol
  - Kent and Canterbury Hospital, Canterbury
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1071005